CLINICAL TRIAL: NCT03296995
Title: Accuracy, Feasibility and Acceptance of Continuous Glucose Monitoring in Critically Systemic Lupus Erythematosus
Brief Title: Accuracy, Feasibility and Acceptance of CGM Lupus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SHRJ001
Record Dates: First submitted 2017-09-25; First posted 2017-09-29 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Systemic Lupus Erythematosus; Critical Illness; Diabetic Blood Glucose Monitoring
Keywords: glucose; systemic lupus erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- flash glucose monitoring system (Experimental): Subjects in the arm measure blood glucose by flash glucose monitoring system.
  Interventions: Device: Flash glucose monitoring system

INTERVENTIONS:
Device: Flash glucose monitoring system — Flash glucose monitoring systems in critically ill patients may improve glycemic control and reduce glucose variability.

SUMMARY:
This is a prospective monocenter, non-randomised, open-lable single-group intervention diagnostic trial on the accuracy, reliability and feasibility of the continuous glucose monitoring system in critically systemic lupus erythematosus (SLE). Newly developed technologies for continuous glucose monitoring in critically SLE patients may improve glycemic control and reduce glucose variability. Critically SLE patients will be performed by continuous glucose monitoring. The subcutaneous glucose will be continuously monitored in critical SLE patients by freestyle libre glucose monitoring system for 14 days. The aim of this study is to evaluate accuracy feasibility and acceptance of these methods. To analyze accuracy sensor glucose levels will be validated due to venous blood measurements with glucose oxidase methods. The influence of several factors like oedema, perspiration, BMI, body temperature, pH-value application of vasoconstrictors on accuracy and feasibility of the particular system would be evaluated. Furthermore the acceptance of physicians and Nursing staff would be evaluated by a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Systemic lupus erythematosus (SLE), as defined by meeting at least 4 of 11 classification criteria of American College of Rheumatology for the classification of systemic lupus erythematosus, either sequentially or coincidentally. The 4 criteria doesn't need to be present at the time of study enrollment;
* critically SLE patients
* informed consent by the patients or legal proxy

Exclusion Criteria:

* age < 18
* no informed consent by the patients or legal proxy
* pregnancy
* infaust prognosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2019-10-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of continuous glucose monitoring compared to glucose oxidase method | 7 d
  Difference between glucose values of continuous glucose monitoring and blood gas analyses

SECONDARY OUTCOMES:
Feasibility of continuous glucose monitoring | 7 d
  Problems within the application of sensor and monitoring during ward routine
Acceptance of continuous glucose monitoring by physicians and nursing staff | 7 d
  Acceptance and evaluation of the device by physicians and nursing staff evaluated by questionnaire

OTHER OUTCOMES:
Technical problems with the monitoring | 7 d
  Number of needed sensors per patient. Duration of functional sensor. Number and reasons for accidentally sensor removal.

CONTACTS AND LOCATIONS:
Locations (1):
- Shuang Ye, MD, Shanghai, Shanghai Municipality, China